CLINICAL TRIAL: NCT05054049
Title: Point of Care Testing (POCT) for Advanced Practitioners (Paramedics) in Urgent and Emergency Care: a Single Site Feasibility Study
Brief Title: Point of Care Testing for Advanced Practitioners (Paramedics)
Acronym: POCTPara
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yorkshire Ambulance Service NHS Trust (Other Government)
Collaborators: University of Bradford (Other)
Responsible Party: Principal Investigator, Dr Fiona Bell, Head of Research & Development, Yorkshire Ambulance Service NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: YASRD148
Record Dates: First submitted 2021-08-06; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Point of Care Testing; Clinical Decision-Making; Community Urgent & Emergency Care; Allied Health Professional
Keywords: Point of Care Testing; Clinical Decision Making; Paramedic; Community Urgent & Emergency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Single site feasibility study
Who Masked: Participant
Masking Description: Patient is randomised to control or intervention arm after consent obtained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abbott i-stat Allinity (Experimental): Randomised patients to this arm receive the application of the point of care testing device to provide further diagnostic information to assist clinical decision making.
  Interventions: Device: Interventional Diagnostic Device Arm
- Usual Care (Placebo Comparator): Randomised patients to this arm receive usual care.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Interventional Diagnostic Device Arm — Point of care testing venous blood diagnostic device.
  Other Names: Abbott i-stat Allinity
  Arms: Abbott i-stat Allinity
Other: Usual care — Usual care provided to patient without use of point of care testing device
  Arms: Usual Care

SUMMARY:
Point of care testing (POCT) is described as a laboratory test conducted near the patient with a rapid result obtained through a portable analysing device, as opposed to the collection of a blood sample being transferred to a central laboratory for analysis and reporting.

Over the past 15 years increasing emphasis has been placed upon the paramedic profession as a possible solution to addressing the increasing demands placed on emergency departments. This is largely viewed through the ability of paramedics to assess patients calling 999 and manage a patient's condition away from the emergency department, with sufficient evidence supporting the role of the paramedic to develop competencies to manage larger volumes of patients.

This feasibility study will seek to understand whether paramedics report that the use of POCT devices is useful in safe clinical decision making with patients in the community, and if it is possible to use the Abbott i-STAT device in the urgent and emergency care setting for those patients where management within the community is being considered.

Given that there is very little evidence in this subject area, the research should start to inform the potential for future innovations in paramedic and community practice, and build on the body of evidence regarding POCT by paramedics related to community management.

ELIGIBILITY:
Inclusion Criteria:

- Paramedic Participants

Inclusion criteria:

* HCPC registered paramedics employed as advanced practitioners
* From the selected advanced practitioner team (Sheffield)
* Able to provide informed consent
* Willing to undergo training and to deliver intervention
* Willing to undergo training to participate in study measures and processes
* Willing to take part in the focus group

Patient Participants

Inclusion criteria:

* Adult patients aged 18 years old and over.
* Registered with a GP Surgery in the Sheffield CCG boundary.
* In their normal home environment, care home, nursing home or step up intermediate bed service, experiencing an ambulatory sensitive presentation related to falls, frailty, mild to moderate breathlessness, or non-specific general illness and receiving an ambulance service response from participating advanced practitioners (paramedics).
* Who do not require immediate life-saving intervention/immediate transfer to ED.
* Able to give written consent during the call-out.

Exclusion Criteria:

-

Paramedic Participants:

• Any HCPC registered advanced practitioner (paramedic) who is currently under investigation for fitness to practice.

Patient Participants

* Patients requiring emergency intervention and immediate transfer to hospital.
* Patient does not have mental capacity.
* Clinical presentations that should not have any delayed on scene time, meeting the criteria outlined in the YAS policy for the assessment, conveyance and referral of patients, for example detailing the NEWS2 score and other appropriate clinical screening tools that assist in the decision making regarding the decision to convey or refer for community management.
* Non-English speaking patients.
* End of life care patients.
* Patients residing in prison.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Self-reported impact of using POCT device | 1.5 hours focus group at end of study
  Qualitative focus group data measuring perceived self-reported impact by advanced practitioner (paramedic).

SECONDARY OUTCOMES:
Non-conveyance rate | Through study completion, expected to be 6 months
  Proportion of cases not conveyed to hospital
72 hour re-contact rate | Through study completion, expected to be 6 months
  Proportion of non-conveyed hospital where there was a re-contact to the ambulance service
Type of POCT cartridges used. | During the procedure
  Type of POCT cartridges used.
Number of POCT cartridges used. | During the procedure
  Number of POCT cartridges used.
Number of successful and unsuccessful attempts in using the POCT device. | During the procedure
  Number of successful and unsuccessful attempts in using the POCT device recorded as a measurement of failure rates
Length of time on scene. | immediately after the patient care episode has ended
  Understanding any changes to time spent with patient
Number of patients who receive POCT. | Through study completion, expected to be 6 months
  Descriptive data to understand how many patients were eligible for the POCT device
Patient demographics and presentations where POCT is applied - age, gender, NEWS2 score, clinical condition. | Through study completion, expected to be 6 months
  Descriptive data to understand patient characteristics of those patients enrolled into study
Feasibility of patient randomisation process | Through study completion, expected to be 6 months
  Descriptive data to record number of successful and unsuccessful attempts at randomisation of eligible patients

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hodge, Principal Investigator — Yorkshire Ambulance Service

IPD SHARING:
Plan to Share IPD: No